CLINICAL TRIAL: NCT05847166
Title: A Phase 2/3, Open-Label Study, to Evaluate the Feasibility and Safety of Intravenous [99mTc]Tc-PSMA-T4 in Subjects with Prostate Cancer
Brief Title: A Phase 2/3,PSMA-T4, Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NCBJ Polatom: Narodowe Centrum Badań Jądrowych Polatom (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PSMA-T4_2021
Record Dates: First submitted 2023-02-17; First posted 2023-05-06 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: The expected duration of participation for each subject is approximately 17 weeks. This includes up to 1 week for screening, 4 weeks for diagnostic procedures, and 12 weeks for safety evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort A - lymph node assessment in intermediate risk group (Active Comparator): The patients will undergo [99mTc]Tc-PSMA-T4 multi-SPECT/CT as an additional modality to contrast-enhanced (CE) multiparametric MRI (according to PI-RADS 2.1 protocol), and chest, and abdominal CE computed tomography and technetium-99m-MDP bone scan in unfavorable risk prostate cancer patients.
  Interventions: Radiation: [99mTc]Tc-PSMA-T4
- Cohort B - general assessment (bone and lymph nodes) in high and very high-risk group (Active Comparator): The patients will undergo [99mTc]TcPSMA-T4 multi-SPECT/CT as an additional modality to CE multiparametric MRI (according to PI-RADS 2.1 protocol), chest, abdomen CE computed tomography, and skeletal scintigraphy (technetium-99m-MDP bone scan).
  Interventions: Radiation: [99mTc]Tc-PSMA-T4
- Cohort C - recurrent disease after definitive treatment (radiotherapy or surgery) (Active Comparator): The patients will undergo [99mTc]Tc-PSMA-T4 multi-SPECT/CT as an additional modality to the second confirmatory imaging modality or biopsy in the case of evidence on progressive disease (PSA persistence/recurrence or radiographic evidence of metastatic disease or clinical symptoms suggesting metastatic disease).
  Interventions: Radiation: [99mTc]Tc-PSMA-T4

INTERVENTIONS:
Radiation: [99mTc]Tc-PSMA-T4 — [99mTc]Tc-PSMA-T4 for intravenous administration. The investigational medicinal product is to be prepared directly in a clinic by radiolabeling the radiopharmaceutical kit containing PSMA-T4 as a drug substance with sodium pertechnetate (99mTc) injection. The [99mTc]Tc-PSMA-T4 radiopharmaceutical should be used for targeted radionuclide SPECT imaging in patients with tumors and metastases of prostate cancer. The investigational medicinal product [99mTc]Tc-PSMA-T4 is dedicated for intravenous administration in radioactivity dose (555 - 740 MBq in cohorts A, B, C.

SUMMARY:
The objectives of this study are to evaluate the feasibility and safety of [99mTc]Tc-PSMA-T4 in the diagnosis and treatment planning of prostate cancer.

DETAILED DESCRIPTION:
This is a Phase 2/3, open-label study, with multicohort design that will enroll up to approximately 80 subjects with prostate cancer (60 for cohorts A, B and 20 for cohort C). Cohort A - lymph node assessment in intermediate risk group before the initiation of treatment.

The patients will undergo [99mTc]Tc-PSMA-T4 multi-SPECT/CT as an additional modality to contrast-enhanced (CE) multiparametric MRI (according to PI-RADS 2.1 protocol), and chest, and abdominal CE computed tomography and technetium-99m-MDP bone scan in unfavorable risk prostate cancer patients.

Cohort B - general assessment (bone and lymph nodes) in high and very high-risk group. The patients will undergo [99mTc]Tc-PSMA-T4 multi-SPECT/CT as an additional modality to contrast-enhanced (CE) multiparametric MRI (according to PI-RADS 2.1 protocol), and chest, and abdominal CE computed tomography and technetium-99m-MDP bone scan in unfavorable risk prostate cancer patients.

Cohort C - recurrent disease after definitive treatment (radiotherapy or surgery) The patients will undergo [99mTc]Tc-PSMA-T4 multi-SPECT/CT as an additional modality to the second confirmatory imaging modality or biopsy in the case of evidence on progressive disease (PSA persistence/recurrence or radiographic evidence of metastatic disease or clinical symptoms suggesting metastatic disease).

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older.
2. PS ECOG < 2
3. Prior diagnosis of any type of prostate cancer with a Gleason score (GlS) above 6.
4. Confirmatory prostate biopsy within 12 weeks (time from pathological diagnosis as PCA date of pathological description to the time of signing the patient's informed consent to participate in the study), only for cohorts A and B.
5. Pelvic mpMRI prostate with PIRADS 2.1 score within 12 weeks before screening, only for cohorts A and B.
6. Willingness to participate in this study and to provide written informed consent.

Additional inclusion criteria for each cohort:

Cohort A:

1. Intermediate risk disease as defined by the most up-to-date version of National Comprehensive Cancer Network Guidelines for Prostate Cancer
2. Greater than 10% chance of lymph node involvement assessed using the Memorial Sloan Kettering nomogram for probability of lymph node involvement in prostate cancer patients.
3. CT of the chest, abdomen and pelvis and bone scan within 12 weeks before screening in the unfavorable risk PC subgroup.
4. No prior treatment for prostate cancer.

Cohort B:

1. High or very high-risk disease as defined by the most up-to-date version of National Comprehensive Cancer Network Guidelines for Prostate Cancer
2. CT of the chest, abdomen and pelvis and bone scan within 12 weeks before screening in the unfavorable risk PC subgroup.
3. No prior treatment for prostate cancer.

Cohort C:

Biochemical failure after radical prostatectomy defined as failure of PSA to fall to undetectable levels (PSA persistence) or undetectable PSA after radical prostatectomy with a subsequent detectable PSA that increases on 2 or more determinations (PSA recurrence) OR biochemical failure after definitive radiotherapy based on Phoenix Consensus (a rise by 2 ng/mL or more above the nadir PSA) OR radiographic evidence of metastatic disease without PSA persistence/recurrence OR clinical symptoms suggesting distant metastases (Roach et al.., 2006).

Exclusion Criteria:

1. No histopathological confirmation of prostate cancer.
2. Patients with pacemakers or metal parts that prevent pelvic MRI to confirm the presence of prostate cancer.
3. Abnormal liver function including a significant increase of liver enzymes like: ALAT, ASPAT, alkaline phosphatase (AP) greater than 5x upper limit normal (ULN) and an increase in bilirubin greater than 2x ULN.
4. Renal impairment including eGFR <30 ml / min.
5. Within 6 months before inclusion into the study: myocardial infarction, other cardiac events requiring hospitalization (unstable angina, etc.), cerebrovascular accident, transient ischemic attack, acute stroke, pulmonary embolism or deep vein thrombosis
6. Acute congestive heart failure or severe arrhythmia (like ventricular arrhythmia), second or higher degree atrio-ventricular (AV) heart block.
7. An active infection that the investigator deems sufficient to exclude the patient from the study, including but not limited to urinary tract infections, respiratory tract infections, and diabetic foot infections with osteomyelitis osteomyelitis.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoints | 17 weeks
  Clinical feasibility in each cohort: the diagnostic method will be deemed a feasible approach if at least 80% of participants in each cohort fulfil the criteria of sensitivity (true positive) and specificity (true negative) of PSMA-T4 WB-SPECT/CT - detection all lesions that are pathologically or radiologically confirmed or suspicious in other modalities recommended in a particular clinical situation by international guidelines for prostate cancer diagnosis and treatment ("golden standards" separate for each cohort). Feasibility = (number of patients with true positive and/or true negative without false positive and/or false negative results of PSMA-T4 WB-SPECT/CT x 100%) / all patients. The patients will undergo PSMA-T4 multi-SPECT/CT as an additional modality to contrast-enhanced (CE) multiparametric MRI (according to PI-RADS 2.1 protocol) withadditional chest and abdominal CE computed tomography and[ 99m Tc]Tc-MDP bone scan in unfavorable risk prostate cancer patients.

SECONDARY OUTCOMES:
Secondary Outcome Measures | 17 weeks
  Sensitivity(number of true positives x 100%)/(number of true positives + number of false negatives) Specificity:(number of true negatives x 100%)/(number of true negatives + number of false positives) Positive and negative predictive value: Positive predictive value defined as number of true positives x 100%/number of true positives + number of false positives. Negative predictive value defined as number of true negatives x 100%/number of true negatives + number of false negatives. The patients will undergo PSMA-T4 multi-SPECT/CT as an additional modality to contrast-enhanced (CE) multiparametric MRI (according to PI-RADS 2.1 protocol) withadditional chest and abdominal CE computed tomography and[ 99m Tc]Tc-MDP bone scan in unfavorable risk prostate cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Garnuszek, Sponsor, Study Director — NCBJ Polatom
Locations (4):
- Poland (4):
  - Centrum Onkologii im. prof. F. Łukaszczyka, Bydgoszcz, Poland
  - Centralny Szpital Kliniczny Uniwersytetu Medycznego, Lodz, Poland
  - GAMMED Centrum Diagnostyczno-Lecznicze, Warsaw, Poland
  - 4. Wojskowy Szpital Kliniczny z Polikliniką SP ZOZ, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: Yes
Clinical Study Report (CSR)
Supporting Information: CSR
Time Frame: 2024
Access Criteria: After contact and approval of the Sponsor